CLINICAL TRIAL: NCT05627882
Title: Evaluation of the Impact of a Forward Viewing Scope at Time of ERCP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Marvin Ryou, Director of Endoscopic Innovations, Brigham and Women's Hospital
Other Study IDs: 2022A002001
Record Dates: First submitted 2022-11-02; First posted 2022-11-28 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Gastro-Intestinal Disorder
Keywords: endoscopy; ERCP
MeSH Terms: conditions — Digestive System Diseases

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Standard ERCP: Patients undergoing ERCP with standard side viewing scope
  Interventions: Diagnostic Test: Forward viewing endoscope

INTERVENTIONS:
Diagnostic Test: Forward viewing endoscope — Additional examination with standard forward viewing endoscope

SUMMARY:
This study will be a prospective, tandem-designed study to determine the proportion of clinically significant missed lesions when using a side- or oblique-viewing endoscope as compared to the standard forward-viewing endoscope. Utilizing standard endoscopy protocols in current practice at Brigham and Women's Hospital, consecutive adult patients undergoing ERCP for traditional reasons will undergo back-to-back tandem EGD and ERCP examinations. This process entails an EGD performed by an attending gastroenterologist first. Next, a second blinded attending gastroenterologist will perform ERCP immediately after index EGD. Both endoscopists will note any clinically significant findings, independent of the other providers procedural findings. Clinically significant findings defined as endoscopic findings that alter patient management (i.e., esophageal varices, peptic ulcer disease, hemorrhage, mass, etc.) during EGD and ERCP will be recorded. As previously stated, some institutions already routinely perform EGD with every ERCP.

DETAILED DESCRIPTION:
BACKGROUND: Endoscopic retrograde cholangiopancreatography (ERCP) is the current procedure of choice for the treatment for a variety of biliary and pancreatic disorders with over 500,000 procedures performed annually in the United States. While the duodenoscope has a unique side-viewing design in order to provide optimal visualization of the major papilla during the ERCP procedure, the non-forward field of view severely limits a complete endoscopic examination of the esophagus and stomach. As a result, key upper gastrointestinal findings, such as peptic ulcer disease or hemorrhage, may be missed given the non-forward viewing design. In a previous retrospective study, significant gastrointestinal findings were not visualized during ERCP with a side-viewing duodenoscope among 19.2% of patients. Given the high miss rate associated with ERCP, performing an esophagogastroduodenoscopy (EGD) with a forward-viewing endoscope may increase the yield of upper gastrointestinal lesions and improve overall patient care. Some centers already routinely employ simultaneous EGD/ERCP.

SPECIFIC AIMS AND OBJECTIVES: The primary aim of this study is to determine the miss rate associated with traditional ERCP. This will be done by supplementing a forward-viewing EGD exam to the traditional side-viewing ERCP procedure. Additionally, the investigators aim to identify patient characteristics associated with clinically significant findings with simultaneous EGD/ERCP. The investigators hypothesize that simultaneous EGD during ERCP will discover clinically significant findings missed by ERCP alone.

STUDY DESIGN: This study will be a prospective, tandem-designed study to determine the proportion of clinically significant missed lesions when using a side- or oblique-viewing endoscope as compared to the standard forward-viewing endoscope. Utilizing standard endoscopy protocols in current practice at Brigham and Women's Hospital, consecutive adult patients undergoing ERCP for traditional reasons will undergo back-to-back tandem EGD and ERCP examinations. This process entails an EGD performed by an attending gastroenterologist first. Next, a second blinded attending gastroenterologist will perform ERCP immediately after index EGD. Both endoscopists will note any clinically significant findings, independent of the other providers procedural findings. Clinically significant findings defined as endoscopic findings that alter patient management (i.e., esophageal varices, peptic ulcer disease, hemorrhage, mass, etc.) during EGD and ERCP will be recorded. As previously stated, some institutions already routinely perform EGD with every ERCP.

STUDY PARTICIPANT SELECTION: Study participants will be selected from the current list of patients undergoing conventional ERCP at Brigham and Women's Hospital. All patients must have a standard indication for the ERCP procedure (i.e., benign or malignant biliary obstruction, choledocholithiasis, etc.) and undergo ERCP with general anesthesia using a conventional duodenoscope to complete the ERCP procedure. Patients undergoing more than one procedure will be eligible to be included in this study for each ERCP procedure. Patients will be recruited from multiple sources including outpatient and inpatient settings or referred from gastrointestinal, oncologic, or primary care providers. Upon arrival, patients will be approached about the study by the advanced endoscopy fellow, study coordinator, attending physician, or member of the gastrointestinal team. Once identified and consented, patients will undergo initial EGD (with a conventional EGD scope) followed by tandem ERCP as described above. To ensure adequate enrollment, a power calculation was performed. Assuming a 19% miss rate1 and 80% power, 144 patients will be required to detect a significant risk difference. To then assess for clinically significant predictors of positive findings, enrollment is estimated to include approximately 500 patients.

STATISTICAL ANALYSIS: For the two comparison groups (EGD findings versus ERCP findings), continuous data will be compared using the two-sample t-test or Wilcoxon rank-sum test and categorical data to be compared using the Chi-square or Fisher's exact test, as appropriate. Multivariable analyses will also be performed using logistic regression to determine significant predictors of missed findings (i.e., patient characteristics) and will be reported as standardized β coefficients as well as odds ratio (OR) with corresponding 95% confidence intervals (CIs). Statistical significance will be defined as a two-tailed P value <0.05. Statistical analyses will be performed using the Stata 15.0 software package (Stata Corp LP, College Station, TX).

ELIGIBILITY:
Inclusion Criteria:

* All adult patients referred for clinically-indicated ERCP

Exclusion Criteria:

* inability to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are referred for clinically indicated ERCP procedure
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-10-14 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with clinically significant endoscopic findings | Intra-procedural
  Endoscopic findings that alter medical/procedural management including: erosive disease, Barrett's esophagus, peptic ulcer, gastrointestinal malignancy, other.

SECONDARY OUTCOMES:
Number of Participants with non-clinically significant endoscopic findings | Intra-procedural
  Endoscopic findings that do not alter medical/procedural management including: gastritis, diverticulum, and hiatal hernia

CONTACTS AND LOCATIONS:
Overall Officials: Marvin Ryou, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Peery AF, Crockett SD, Murphy CC, Lund JL, Dellon ES, Williams JL, Jensen ET, Shaheen NJ, Barritt AS, Lieber SR, Kochar B, Barnes EL, Fan YC, Pate V, Galanko J, Baron TH, Sandler RS. Burden and Cost of Gastrointestinal, Liver, and Pancreatic Diseases in the United States: Update 2018. Gastroenterology. 2019 Jan;156(1):254-272.e11. doi: 10.1053/j.gastro.2018.08.063. Epub 2018 Oct 10. PMID 30315778
- [Background] Thomas A, Vamadevan AS, Slattery E, Sejpal DV, Trindade AJ. Performing forward-viewing endoscopy at time of pancreaticobiliary EUS and ERCP may detect additional upper gastrointestinal lesions. Endosc Int Open. 2016 Feb;4(2):E193-7. doi: 10.1055/s-0041-109084. Epub 2016 Jan 11. PMID 26878048
- [Background] Ford AC, Marwaha A, Lim A, Moayyedi P. What is the prevalence of clinically significant endoscopic findings in subjects with dyspepsia? Systematic review and meta-analysis. Clin Gastroenterol Hepatol. 2010 Oct;8(10):830-7, 837.e1-2. doi: 10.1016/j.cgh.2010.05.031. Epub 2010 Jun 10. PMID 20541625